CLINICAL TRIAL: NCT02533414
Title: Effect of Use of Ureteral Access Sheath on Blood and Urine Levels of Netrin-1 in Patients Undergoing Retrograde Intrarenal Surgery
Brief Title: Effect of Use of Ureteral Access Sheath on Levels of Netrin-1 in Patients Undergoing RIRS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Selcuk University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Ozcan Kilic, Associate Professor, M.D., Selcuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SU-RIRS-UAS-04
Record Dates: First submitted 2015-08-23; First posted 2015-08-26 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-03

CONDITIONS: Urolithiasis
Keywords: kidney stone; retrograde intrarenal surgery; ureteral access sheath; kidney function
MeSH Terms: conditions — Urolithiasis; Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UAS (+) (Experimental): RIRS with UAS: A ureteral access sheath (UAS) will be positioned into the ureter of the patient prior to the insertion of the flexible ureterorenoscope (RIRS).
  Interventions: Device: RIRS with UAS
- UAS (-) (Active Comparator): RIRS without UAS: A ureteral access sheath (UAS) will not be positioned into the ureter of the patient prior to the insertion of the flexible ureterorenoscope (RIRS).
  Interventions: Device: RIRS without UAS

INTERVENTIONS:
Device: RIRS with UAS — Ureteral access sheath (UAS) will be used during RIRS.
  Arms: UAS (+)
Device: RIRS without UAS — Ureteral access sheath will not be used during RIRS.
  Arms: UAS (-)

SUMMARY:
In this study, it is aimed to evaluate whether use of a ureteral access sheath (UAS) during retrograde intrarenal surgery (RIRS) due to kidney stone has any effect on protecting the kidney functions by measuring blood and urine and Netrin-1 levels.

DETAILED DESCRIPTION:
This study will include patients aged between 18 and 65 who will undergo retrograde intrarenal surgery (RIRS) due to renal stone(s). A total of 60 patients (male or female) will be recruited, and will be randomized into 2 groups consisting of 30 patients in each group. The first group of patients will undergo RIRS with a ureteral access sheath (UAS) positioned prior to surgery; and the second group will undergo RIRS without UAS. As use of UAS decreases the pressure in the renal pelvis during RIRS, it is aimed to evaluate whether using UAS or not affects the kidney functions. Besides the routine kidney function tests, namely urea and creatinine, and Netrin-1 (more specific and early marker of kidney function) will be used to assess the differences in the kidney functions. Preoperative blood urea, creatinine and Netrin-1 levels and urine Netrin-1 levels will be studied for all patients. After the surgery, blood urea and creatinine levels will be again studied as well as blood Netrin-1 levels at postoperative 48th hour; and urine Netrin-1 levels at postoperative 24th hour.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18-65 years old
* Having an indication of retrograde infrarenal surgery (RIRS) due to kidney stone

Exclusion Criteria:

* Patients with uncontrolled diabetes mellitus and diabetic nephropathy
* Patients with blood pressure > 140/80 mmHg despite regular use of antihypertensive agent(s)
* Patients with chronic kidney failure who need dialysis
* Patients who have had prerenal, renal or postrenal acute kidney failure 3 months or much earlier
* Patients who have had pyelonephritis 3 months or much earlier
* Patients younger than 18 years or older than 65 years
* Patients who have undergone a kidney surgery within the last 3 months and have abnormal kidney function tests
* Patients with a concomitant ureter stone who will undergo an endoscopic ureter stone treatment at the same session

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-08 (Actual); Primary Completion 2017-06 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Blood Netrin-1 level (pg/mL) | Within the first 48 hours after the surgery (RIRS)
  Determination of any impairment in renal function when ureteral access sheath is not used during RIRS by measuring blood Netrin-1 level.

SECONDARY OUTCOMES:
Urine Netrin-1 level (pg/mL) | Within the first 24 hours after the surgery (RIRS)
  Determination of any impairment in renal function when ureteral access sheath is not used during RIRS by measuring urine Netrin-1 level.
Blood urea level (mg/dL) | Within the first 7 days after surgery (RIRS)
  Determination of any impairment in renal function when ureteral access sheath is not used during RIRS by measuring blood urea levels.
Blood creatinine level (mg/dL) | Within the first 7 days after surgery (RIRS)
  Determination of any impairment in renal function when ureteral access sheath is not used during RIRS by measuring blood creatinine levels.

CONTACTS AND LOCATIONS:
Overall Officials: Ozcan Kilic, MD, Principal Investigator — Selcuk University, School of Medicine, Department of Urology
Locations (1):
- Selcuk University, School of Medicine, Department of Urology, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cepeda M, Amon JH, Mainez JA, Rodriguez V, Alonso D, Martinez-Sagarra JM. Flexible ureteroscopy for renal stones. Actas Urol Esp. 2014 Nov;38(9):571-5. doi: 10.1016/j.acuro.2014.03.014. Epub 2014 Jun 2. English, Spanish. PMID 24881777
- [Background] Oguz U, Resorlu B, Ozyuvali E, Bozkurt OF, Senocak C, Unsal A. Categorizing intraoperative complications of retrograde intrarenal surgery. Urol Int. 2014;92(2):164-8. doi: 10.1159/000354623. Epub 2014 Feb 6. PMID 24503707
- [Background] Aboumarzouk OM, Monga M, Kata SG, Traxer O, Somani BK. Flexible ureteroscopy and laser lithotripsy for stones >2 cm: a systematic review and meta-analysis. J Endourol. 2012 Oct;26(10):1257-63. doi: 10.1089/end.2012.0217. Epub 2012 Jul 30. PMID 22642568
- [Background] Auge BK, Pietrow PK, Lallas CD, Raj GV, Santa-Cruz RW, Preminger GM. Ureteral access sheath provides protection against elevated renal pressures during routine flexible ureteroscopic stone manipulation. J Endourol. 2004 Feb;18(1):33-6. doi: 10.1089/089277904322836631. PMID 15006050
- [Background] Kourambas J, Byrne RR, Preminger GM. Does a ureteral access sheath facilitate ureteroscopy? J Urol. 2001 Mar;165(3):789-93. PMID 11176469
- [Background] L'esperance JO, Ekeruo WO, Scales CD Jr, Marguet CG, Springhart WP, Maloney ME, Albala DM, Preminger GM. Effect of ureteral access sheath on stone-free rates in patients undergoing ureteroscopic management of renal calculi. Urology. 2005 Aug;66(2):252-5. doi: 10.1016/j.urology.2005.03.019. PMID 16040093
- [Background] Stern JM, Yiee J, Park S. Safety and efficacy of ureteral access sheaths. J Endourol. 2007 Feb;21(2):119-23. doi: 10.1089/end.2007.9997. PMID 17338606
- [Background] Traxer O, Wendt-Nordahl G, Sodha H, Rassweiler J, Meretyk S, Tefekli A, Coz F, de la Rosette JJ. Differences in renal stone treatment and outcomes for patients treated either with or without the support of a ureteral access sheath: The Clinical Research Office of the Endourological Society Ureteroscopy Global Study. World J Urol. 2015 Dec;33(12):2137-44. doi: 10.1007/s00345-015-1582-8. Epub 2015 May 14. PMID 25971204
- [Background] Shlipak MG, Mattes MD, Peralta CA. Update on cystatin C: incorporation into clinical practice. Am J Kidney Dis. 2013 Sep;62(3):595-603. doi: 10.1053/j.ajkd.2013.03.027. Epub 2013 May 20. PMID 23701892
- [Background] Delanaye P, Cavalier E, Morel J, Mehdi M, Maillard N, Claisse G, Lambermont B, Dubois BE, Damas P, Krzesinski JM, Lautrette A, Mariat C. Detection of decreased glomerular filtration rate in intensive care units: serum cystatin C versus serum creatinine. BMC Nephrol. 2014 Jan 13;15:9. doi: 10.1186/1471-2369-15-9. PMID 24410757
- [Background] Barallobre MJ, Pascual M, Del Rio JA, Soriano E. The Netrin family of guidance factors: emphasis on Netrin-1 signalling. Brain Res Brain Res Rev. 2005 Jul;49(1):22-47. doi: 10.1016/j.brainresrev.2004.11.003. Epub 2005 Jan 15. PMID 15960985
- [Background] Ramesh G, Krawczeski CD, Woo JG, Wang Y, Devarajan P. Urinary netrin-1 is an early predictive biomarker of acute kidney injury after cardiac surgery. Clin J Am Soc Nephrol. 2010 Mar;5(3):395-401. doi: 10.2215/CJN.05140709. Epub 2009 Dec 10. PMID 20007677